CLINICAL TRIAL: NCT01260805
Title: A Phase I, Open Label, Randomized, Two-Way Crossover, Single Dose Study To Determine The Bioequivalence Of Ethinylestradiol + Gestodene - Harmonet 0,02mg + 0,075mg (Laboratórios Pfizer Ltda.) In The Sugar Coated Tablets Form, Versus Femiane® 0,02mg + 0,075mg (Schering Do Brasil Química E Farmacêutica Ltda.), In The Sugar Coated Tablets Form, Under Fasted Conditions In Female And Healthy Volunteers.
Brief Title: A Bioequivalence Study Of Ethinylestradiol + Gestodene In Female And Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B3341001; ICF PBIO 071/10 APH 100214
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Bioequivalence; Ethinylestradiol; Gestodene; Harmonet
Keywords: bioequivalence; study; ethinylestradiol; gestodene
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference Drug (Active Comparator)
  Interventions: Drug: Reference Drug
- Test Drug (Active Comparator)
  Interventions: Drug: Test Drug

INTERVENTIONS:
Drug: Reference Drug — Femiane® Ethinylestradiol 0,02mg + Gestodene 0,075mg sugar coated tablets single dose
  Arms: Reference Drug
Drug: Test Drug — Harmonet® Ethinylestradiol 0,02mg + Gestodene 0,075mg sugar coated tablets single dose
  Arms: Test Drug

SUMMARY:
A Phase I, Open Label, Randomized, Two-way Crossover, Single Dose Study to Determine the Bioequivalence of Ethinylestradiol + Gestodene - The objective of the study is to verify through a single dose study, if the two formulations of Ethinylestradiol 0,02mg + Gestodene 0,075mg sugar coated tablets are bioequivalent when administered at the same dose and under fasting conditions.

DETAILED DESCRIPTION:
Bioequivalence Study

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects in childbearing age, between the ages of 18 and 45 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* The BMI - Body Mass Index of the volunteers should be within the range of 18,5 to 24,9 (Dietary Guidelines for Americans) and it may vary up to 10% due to the upper limit (18,5 to 27,39) and total body weight >50kg
* Do not be a smoker (at least 3 months);
* Not be using hormone contraceptives for at least 28 days before the medication dosing;
* Women with a regular menstrual cycle (menstrual cycle that occurs, in average, in each 28 days, varying from 25 to 35 days);
* Use lubricated condoms with spermicidal or diaphragm with spermicidal (in accordance with the volunteer's preference)
* Systolic Pressure up to 130mmHg;
* Diastolic Pressure up to 85mmHg;
* An informed consent document signed and dated by the subject or a legally acceptable representative. If the subject and/or legally acceptable representative cannot read, then the informed consent document may be signed by an impartial witness.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* The volunteer has a drug abuse history [subjects using marijuana and hashish will be excluded if they have used these drugs less than three months prior to the medical consult and for drugs such as cocaine, phencyclidine (PCP), crack and heroin, volunteers will be excluded that have used these drugs less than 1 year prior to the medical consult.
* A positive exam for drugs in urine (Methamphetamine, Opiate, Morphine, Marijuana, Cannabis, Amphetamine, Coccaine, Benzoylecgogine, Benzodiazepine) or a positive test for alcohol before the internment in periods 1 and 2.
* History of regular alcohol consumption exceeding 7 drinks/week (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor) within 6 months of screening.
* The volunteer is a smoker or having stopped smoking less than 3 months
* The volunteer has participated of any experimental trial or has ingested any experimental drug within the 6 months that precede the beginning of the study (ANVISA: Resolution RDC nº34, from June 3rd 2008).
* 12-lead ECG demonstrating QTc >450 msec at screening. If QTc exceeds 450 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility.
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of non-hormonal contraception as outlined in this protocol from at least 14 days prior to the first dose of study medication.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal medicine, herbal supplements must be discontinued 28 days prior to the first dose of study medication. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
* Hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing IUDs, postcoital contraceptive methods) and hormone replacement therapy must be discontinued 28 days prior to the first dose of study medication.
* Implant (ex. Norplant®) or a progesterone depot injection (ex. Depo-Provera®) or the use of any dispositive for the long term treatment with progesterone or estrogens (ex. Estring®) up to 6 months before the administration of the medication in study;
* A depot injection or an implant of any active ingredient up to 3 months before the administration of the medication in study;
* Have used an injection contraceptive of Medroxyprogesterone Acetate one year before the beginning of the study;
* Have had sexual intercourse without a contraceptive method (preservative, IUD, diaphragm with spermicidal) within the last 14 days.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Maxium concentration (Cmax) for ethinylestradiol/gestodene in plasma | Up to 96h / Up to 144h
Area under the plasma/serum/blood concentration(AUC0-t) time curve from time zero to time t for ethinylestradiol/gestodene | Up to 96h / Up to 144h

SECONDARY OUTCOMES:
Area under the curve (AUC0-inf) for ethinylestradiol/gestodene | Up to 96h / Up to 144h
Time of maximum concentration (Tmax) for ethinylestradiol/gestodene in plasma | Up to 96h / Up to 144h
Elimination of half-life(T1/2) for ethinylestradiol/gestodene | Up to 96h / Up to 144h
K el for ethinylestradiol/gestodene | Up to 96h / Up to 144h
Area under the curve from the time of dosing (AUC t/inf) extrapolated to infinity for ethinylestradiol/gestodene | Up to 96h / Up to 144h

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Aparecida de Goiânia, Goiás, Brazil

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3341001&StudyName=A%20Bioequivalence%20Study%20Of%20Ethinylestradiol%20+%20Gestodene%20In%20Female%20And%20Healthy%20Volunteers.